CLINICAL TRIAL: NCT06212596
Title: A Randomised Phase II Trial of Selinexor, Cyclophosphamide and Prednisone vs Cyclophosphamide and Prednisone in Relapsed or Refractory Multiple Myeloma (RRMM) Patients
Brief Title: Selinexor, Cyclophosphamide and Prednisone in Myeloma
Acronym: MUKtwelve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM17/95228; 2017-001736-19 (EudraCT Number)
Record Dates: First submitted 2017-06-14; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — selinexor; Cyclophosphamide; Prednisone

STUDY DESIGN:
Intervention Model Description: Participants will be randomised on a 3:1 basis to receive either selinexor + cyclophosphamide + prednisone (SCP) or cyclophosphamide + prednisone (CP). A computer-generated minimisation programme that incorporates a random element will be used to ensure treatment groups are well-balanced for pre-specified factors:
  * Age (<60 vs. 60-69 years vs. ≥70 years )
  * Number of prior lines of therapy (≤3 vs. >3)
  A maximum of 60 participants will be recruited (45 participants in the SCP arm, and 15 participants in the CP arm).
  Participants who experience disease progression on the CP arm, may receive SCP, once progression has been confirmed by the CTRU and the participant has been deemed eligible to receive SCP. Patients randomised to SCP have no further trial treatment stipulated following SCP therapy. The analysis of the treatment switch phase of the trial is exploratory.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selinexor cylophosphamide prednisone (Experimental): Participants will receive treatment with Selinexor, Cyclophosphamide and Prednisone.
  Interventions: Drug: Selinexor; Drug: Cyclophosphamide; Drug: Prednisone
- Cyclophosphamide predinisone (Active Comparator): Participants will receive treatment with Cyclophosphamide and Prednisone. Participants who experience disease progression on the CP arm, may receive SCP.
  Interventions: Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: Selinexor — Selinexor is a Selective Inhibitor of Nuclear Export (SINE) compound that binds and inactivates Exportin 1 (XPO1), thereby forcing the nuclear retention of key tumour suppressor proteins (TSPs). Selinexor is an oral, first-in-class, potent, slowly reversible, covalent-binding Selective Inhibitor of Nuclear Export (SINE) compound that specifically blocks the karyopherin protein Exportin 1 (XPO1), also called chromosome region maintenance 1.
  Arms: Selinexor cylophosphamide prednisone
Drug: Cyclophosphamide — Cyclophosphamide is a long used conventional chemotherapy with potent anti-myeloma activity and low toxicity when administered at low doses as in the current protocol (Hajek et al. (2016)). It is being extensively used in combination with novel agents, including bortezomib, lenalidomide, and pomalidomide, and provides a cost-effective and well-tolerated alternative as a combination partner (Morgan et al. (2007); Mai et al. (2015); Baz et al. (2016)).
Drug: Prednisone — Steroids have been a very effective backbone for every myeloma combination therapy developed so far. Prednisone is the standard steroid in a number of widely used regimens (Mateos et al. (2010);Palumbo et al. (2006)). Decreasing the morbidity associated with high dose steroid use by using better-tolerated regimens addresses a large unmet need of the myeloma patient population.

SUMMARY:
The trial is designed as a randomised, controlled, open, parallel group, multi-centre phase II trial to evaluate clinical efficacy of selinexor in combination with cyclophosphamide and prednisone.

DETAILED DESCRIPTION:
The trial is designed as a randomised, controlled, open, parallel group, multi-centre phase II trial to evaluate clinical efficacy of selinexor in combination with cyclophosphamide and prednisone. Selinexor is the first-in-class selective inhibitor of nuclear export (SINE). Selinexor forms slowly reversible adducts with the substrate binding pocket of Exportin and has been demonstrated to lead to effective cell kill by causing accumulation pro-apoptotic proteins in the nucleus of myeloma cells. To maximise response to this novel drug in a relapsed-refractory setting, Selinexor will be combined with low-dose cyclophosphamide and prednisone. Lower, continuous doses of cyclophosphamide and intermittent doses of prednisone have been chosen to limit toxicity for the triplet regimen in the elderly myeloma patient population. A calibration group will receive cyclophosphamide plus prednisone alone, and will be used to evaluate the validity of the outcome in the experimental group.

Participants will be randomised on a 3:1 basis to receive either selinexor + cyclophosphamide + prednisone (SCP) or cyclophosphamide + prednisone (CP).

A maximum of 60 participants will be recruited (45 participants in the SCP arm, and 15 participants in the CP arm).

Participants who experience disease progression on the CP arm, may receive SCP, once progression has been confirmed by the CTRU and the participant has been deemed eligible to receive SCP. Patients randomised to SCP have no further trial treatment stipulated following SCP therapy. The analysis of the treatment switch phase of the trial is exploratory.

Participants will be recruited from approximately 10 NHS Hospitals throughout the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent and willing to follow all trial protocol assessments
2. Aged 18 years or over
3. Participants with confirmed myeloma based on International Myeloma Working Group (IMWG) criteria (Rajkumar et al. (2014))
4. Measurable disease with at least one of the following:

   * Paraprotein ≥5g/L
   * Serum free light chains ≥100mg/L with abnormal ratio for light chain only myeloma
   * Bence Jones protein ≥200mg/L
5. Participants with relapsed or relapsed refractory myeloma who have received ≥ 2 prior anti-myeloma treatments including a proteasome inhibitor and lenalidomide, and now require further treatment
6. Patients for which cyclophosphamide and prednisone alone would be a suitable treatment
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
8. Female participants of childbearing potential must agree to use two methods of contraception (including one highly effective and one effective method of contraception) and have a negative urine pregnancy test at screening.

   Male participants must use an effective barrier method of contraception if sexually active with a female of childbearing potential.

   For both male and female participants, effective methods of contraception must be used throughout the trial and for at least 36 months following the last dose of trial treatment
9. Required laboratory values within 14 days prior to randomisation:

   * Platelet count ≥50x109/L. Platelet count of 30-50 is acceptable if bone marrow aspirate or trephine shows tumour replacement of >50%. Platelet support is permitted within 14 days prior to randomisation, although platelet transfusions to help participants meet eligibility criteria are not allowed within 72 hours prior to the blood sample to confirm protocol eligibility
   * Absolute neutrophil count ≥1.0 x 109/L. Growth factor support is not permitted within 14 days prior to randomisation
   * Haemoglobin ≥ 8090 g/L. Blood support is permitted
   * Alanine transaminase (ALT) and / or aspartate transaminase (AST) ≤3 x upper limit of normal
   * Creatinine clearance ≥ 2030 ml/min (using Cockcroft Gault formula)
   * Bilirubin ≤1.5 x upper limit of normal . Gilberts syndrome patients must have a total bilirubin ≤3 x upper limit of normal

Exclusion Criteria:

1. The following participants will be excluded:

   * those with non-measurable disease
   * those with a solitary bone or solitary extramedullary plasmacytoma
   * plasma cell leukaemia
2. Participants with a history of malignancy (other than myeloma) within 5 years before the date of randomisation (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that, in the opinion of the investigator, with concurrence with the Chief Investigator, is considered cured with minimal risk of recurrence within 5 years)
3. Participants with a known or underlying uncontrolled concurrent illness that, in the investigator's opinion, would make the administration of the trial drug hazardous or circumstances that could limit compliance with the trial, including, but not limited to the following:

   * acute or chronic graft versus host disease
   * uncontrolled hypertension
   * symptomatic congestive heart failure
   * unstable angina pectoris
   * myocardial infarction within past 6 months
   * uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4 GradeCTCAE grade ≥2)
   * active symptomatic fungal, bacterial, and/or viral infection including known active HIV or known viral (A, B or C) hepatitis
   * psychiatric or social conditions that may interfere with participant compliance
   * uncontrolled (i.e., clinically unstable) infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; however, prophylactic use of these agents is acceptable even if parenteral
   * or any other condition (including laboratory abnormalities) that in the opinion of the Investigator places the participant at unacceptable risk for adverse outcome if he/she were to participate in the trial
4. Participants who have previously received Selinexor or any other SINE compound
5. Previous anti-tumour therapies including investigational medicinal products at any dose within 28 days before the start of protocol treatment.

   * Prednisone up to a dose of 175 mg per week may be given between screening and the beginning of treatment if medically required but should be stopped before trial treatment starts.
   * Bisphosphonates for bone disease are also permitted
6. Participants with a history of a refractory nausea, diarrhoea, vomiting, malabsorption, gastrointestinal surgery or other procedures or conditions that might, in the opinion of the Investigator, interfere with the absorption or swallowing of the trial drug(s)
7. Peripheral neuropathy of CTCAE grade ≥ grade 32 (or ≥ grade 21 with pain) severity (as per NCI-CTCAEv4.0 )
8. Female participants who are lactating or have a positive pregnancy test at screening
9. Known allergy or previous intolerance to any of the trial medications, their analogues, or excipients in the various formulations of any agent that would prevent the participant receiving these as directed in the protocol
10. Major surgery within 14 days prior to randomisation
11. Radiotherapy within 7 days prior to randomisation for palliative pain control or therapeutic radiotherapy within 14 days prior to randomisation
12. Chemotherapy or immunotherapy or any other anticancer therapy within 2 weeks prior to Cycle 1 Day 1 or radio-immunotherapy 4 weeks prior to Cycle 1 Day 1 (NB: except steroids in the doses outlined above)
13. Myeloma involving the Central Nervous System

SCP following CP Inclusion Criteria

1. Randomised to CP on the MUKtwelve trial, has tolerated treatment and can continue on CP during the SCP treatment, and received at least one full cycle of treatment
2. Centrally confirmed disease progression by IMWG criteria. This must be confirmed by two consecutive assessments based on local lab results. Local laboratory reports must be sent to CTRU to confirm progression and site must have received confirmation of progression from CTRU.
3. ECOG performance status ≤2
4. Required laboratory values within 14 days prior to starting treatment on SCP:

   * Platelet count ≥50x109/L. Platelet count of 30-50 is acceptable if bone marrow aspirate or trephine shows tumour replacement of >50%. Platelet support is permitted within 14 days prior to starting SCP, although platelet transfusions to help participants meet eligibility criteria are not allowed within 72 hours prior to the blood sample to confirm protocol eligibility
   * Absolute neutrophil count ≥1.0 x 109/L.
   * Haemoglobin ≥ 80 g/L. Blood support is permitted
   * Alanine transaminase (ALT) and / or aspartate transaminase (AST) ≤3 x upper limit of normal
   * Creatinine clearance ≥ 20 ml/min (using Cockcroft Gault formula)
   * Bilirubin ≤1.5 x upper limit of normal. Suspected Gilberts syndrome patients must have a total bilirubin ≤3 x upper limit of normal
   * B2M
5. Female participants of childbearing potential must agree to use two methods of contraception (including one highly effective and one effective method of contraception) and have a negative urine pregnancy test at screening.

Male participants must use an effective barrier method of contraception if sexually active with a female of childbearing potential.

For both male and female participants, effective methods of contraception must be used throughout the trial and for 12 months following the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 6 months | 6 months
  To determine whether the addition of selinexor to cyclophosphamide and prednisone may lead to an increased progression free survival

SECONDARY OUTCOMES:
Number of SAEs, SARs, SUSARs | 3 1/2 years
  Safety will be reported based on the number of safety events seen
Progression free survival | 6 and 12 months
  Progression-free survival is defined as the time from randomisation to first documented evidence of disease progression or death. Participants who have not progressed at the time of analysis will be censored at the last date they were known to be alive and progression-free.
Maximum response | 6 and 12 months
  Response to treatment is assessed as per the Modified IWG Uniform Response Criteria given in Appendix 1. Maximum response is defined as the proportion of participants achieving each of the response categories sCR, CR, VGPR, PR, MR or SD as their maximum response to treatment. Participants who do not have at least one post-baseline response assessment will be excluded from the analysis of this endpoint.
Time to maximum response | 6 and 12 months
  Time to maximum response is defined as the time from randomisation until the participant achieves any of the categories sCR, CR, VGPR, PR, MR or SD as their maximum response. Participants who do not achieve a maximum response will either be classed as having had a competing risk or censored at the time of disease progression or death, whichever is earlier
Duration of response | 6 and 12 months
  Response duration is defined as the time from the first observation of at least PR until disease progression. Participants who die due to causes other than progression will be censored at the time of death. Participants who, at the time of analysis, have not progressed, will be censored at the date last known to be alive and progression-free. Participants not achieving at least a PR are not included in this analysis.
Compliance to therapy | 6 months
  Compliance to therapy will be summarised by mean dose, number of doses missed and number of dose reductions and delays throughout the treatment period. The reasons for missed and dose modifications will also be summarised.
Number of participants with treatment-related adverse events as assessed by CTCAE 4.0 (time frame: 3 ½ years) | 3 1/2 years
  Toxicity analyses will summarise by trial arm and show the proportion of participants experiencing each grade of toxicity overall, and during each treatment cycle. For more detailed summaries, this information will also be broken down into the different types of toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kaiser, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (13):
- United Kingdom (13):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew Hospital, London
  - Guys and St Thomas NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Marsden Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Sheffield Teaching Hospitals NHS Foundation Trust, Northern General Hospital, Sheffield
  - University Hospital Southampton, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Worthing Hospital, Worthing

IPD SHARING:
Plan to Share IPD: No